CLINICAL TRIAL: NCT07291505
Title: Investigation of the Predictability of Kinesiophobia on Functional Outcomes in Conservatively Treated Distal Radius Fractures
Brief Title: The Investigation of Kinesiophobia in Conservative Distal Radius Fractures
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-789644
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Distal Radius Fracture; Kinesiophobia; Functional Status
Keywords: Tampa Scale of Kinesiophobia; distal radius fracture; wrist function; upper extremity weight bearing
MeSH Terms: conditions — Wrist Fractures; Kinesiophobia | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated conservatively with a diagnosis of distal radius fracture
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — A goniometric assessment will be performed to measure the range of motion in the wrist-forearm joint, and a Push Off test will be conducted to measure the upper extremity weight-bearing capacity.
  Additionally, the Tampa Scale of Kinesiophobia and Patient-Rated Wrist Evaluation Questionnaire will be administered to patients using a face-to-face assessment method.

SUMMARY:
This study aimed to investigate the predictability of kinesiophobia on functional outcomes in conservatively treated patients with distal radius fractures. For this purpose, patients' level of kinesiophobia will be assessed using the Tampa Kinesiophobia Scale. To assess the functional status of patients, joint range of motion and upper extremity weight bearing measurements will be performed. Patients' functionality will be additionally assessed with the Patient Rated Wrist Evaluation Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Having been treated conservatively with an isolated distal radius fracture diagnosis,
* Having a cognitive level that allows one to understand assessment methods and apply instructions.

Exclusion Criteria:

* Comorbid musculoskeletal-neurovascular injuries
* Bilateral injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers among the patients who were referred to the hand rehabilitation unit after being followed conservatively with a diagnosis of distal radius fracture in the hand surgery clinic of a university hospital will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia | At 12 and 18 weeks after injury
  It is a 17-item scale scored using a 4-point Likert scale (1 = Strongly disagree, 4 = Strongly agree). A total score is calculated after reversing items 4, 8, 12, and 16. The individual receives a total score between 17 and 68. A high score on the scale indicates a high level of kinesiophobia.
Goniometric measurement | At 12 and 18 weeks after injury
  Patients' forearm pronation and supination, as well as wrist flexion, extension, radial and ulnar deviation movements, will be measured using a universal goniometer.
Push-Off Test | At 12 and 18 weeks after injury
  It determines the force that the person can exert on their injured limb. The measurement will be taken using a Jamar hand dynamometer. While the person is standing, with the shoulder at 30 degrees of extension and the elbow at 30 degrees of flexion, the measurement will be repeated three times and the average recorded in kilograms.
Patient-Rated Wrist Evaluation | At 12 and 18 weeks after injury
  It measures the severity of wrist pain and the level of disability in activities of daily living. The survey consists of two subsections with a total of 15 questions. Each question is answered on a scale of 0 to 10 (0 = no pain/difficulty; 10 = maximum pain felt/inability to perform). The scores for the pain and function sections are added together to determine the final score, which is calculated out of 100. A high score indicates a high level of pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jayakumar P, Teunis T, Vranceanu AM, Lamb S, Ring D, Gwilym S. Early Psychological and Social Factors Explain the Recovery Trajectory After Distal Radial Fracture. J Bone Joint Surg Am. 2020 May 6;102(9):788-795. doi: 10.2106/JBJS.19.00100. PMID 32379119
- [Background] Goudie ST, Broll R, Warwick C, Dixon D, Ring D, McQueen M. The Association Between Psychological Factors and Outcomes After Distal Radius Fracture. J Hand Surg Am. 2022 Feb;47(2):190.e1-190.e10. doi: 10.1016/j.jhsa.2021.04.012. Epub 2021 Jun 8. PMID 34112544